CLINICAL TRIAL: NCT02946229
Title: Data Collection for Next Generation Ultrasound Technology Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 110.04-2016-GES-0005
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Endstage Renal Disease
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: The study is designed to collect data from a ultrasound device being used to evaluate feasibility of next generation algorithms for ultrasound data processing and does not test any health outcome. All eligible adults (aged 18 or older) will contribute case data from a convenience sample of maintenance hemodialysis population available at the study site and consistent with feasibility assessment of the technology. A relatively large feasibility population is used due to the need to test feasibility of multiple features across variations within this population.
Oversight: Data Monitoring Committee: No

ARMS (1):
- MHD Population Ultrasound (Other): Eligible subjects in a convenience population at the site (Maintenance Hemodialysis, MHD) incidentally undergoingnon-invasive cardiac, pulmonary, and abdominal ultrasound scanning on the commercially available GE Vivid S70 system for use in testing feasibility of new algorithms for processing this data.
  Interventions: Device: Ultrasound scan

INTERVENTIONS:
Device: Ultrasound scan — Collection of ultrasound data sets that include routine ultrasound data (eg, extravascular lung fluid, cardiac velocity time integral and inferior vena cava) on the commercial GE Vivid S70 Ultrasound System which are used to test feasibility of next generation ultrasound algorithms being developed to process these data types.

SUMMARY:
The study is designed to collect data from a ultrasound device being used to evaluate feasibility of next generation algorithms for ultrasound data processing and does not test any health outcome.

DETAILED DESCRIPTION:
The study is designed to collect data from a ultrasound device being used to evaluate feasibility of next generation algorithms for ultrasound data processing and does not test any health outcome. All eligible adults (aged 18 or older) will contribute case data from a convenience sample of maintenance hemodialysis population available at the study site and consistent with feasibility assessment of the technology. A relatively large feasibility population is used due to the need to test feasibility of multiple features across variations within this population.

ELIGIBILITY:
Inclusion Criteria:

1. Are adults (aged 18 years of age or older) at the time of consent;
2. Are undergoing maintenance hemodialysis (MHD); AND
3. Are able and willing to provide written informed consent for participation

Exclusion Criteria:

1. Have anatomical characteristics or comorbid medical conditions that prevent completion of ultrasound scanning using the study device; OR
2. Are potentially put at additional risk by participating, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, MD, Principal Investigator — Research By Design, LLC
Locations (1):
- Research By Design, Evergreen Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MHD Population Ultrasound
Started | 142
Completed | 142
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Arm/Group | MHD Population Ultrasound
Number analyzed (Participants) | 142
Age, Customized [Count of Participants; unit: Participants]
  >=18 years | 142
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender information not collected
  Participants
    Male or Female | 142

OUTCOME MEASURES:

1. Primary Outcome: Number of Diagnostic Ultrasound Exams
Description: Collection (number) of ultrasound images representative of sonographic findings routinely observed in the general imaging population.
Time Frame: 1 day
Population: No performance or efficacy data were studied; No statistical analysis was performed per the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | MHD Population Ultrasound
Number analyzed (Participants) | 142
Participants | 142

ADVERSE EVENTS:
Arm/Group | MHD Population Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No